CLINICAL TRIAL: NCT03476343
Title: Clinical Use of a Neonatal MRI System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIN_NICUclinicalMRI_003
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: NICU MRI
Keywords: NICU; MRI; Neonatal; Cincinnati

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MRI for Neonates (Experimental): MRI
  Interventions: Device: GE OPTIMA MR430s with HDx/GE Electronics

INTERVENTIONS:
Device: GE OPTIMA MR430s with HDx/GE Electronics — MRI scan

SUMMARY:
The purpose of the present study is to continue clinical scanning on the NICU MRI with improved administrative processes and procedures, thereby making medically indicated, state of the art/high end MRI exams available to all infants treated at CCHMC.

DETAILED DESCRIPTION:
There are significant safety and image quality issues associated with transferring neonates from the Neonatal Intensive Care Unit (NICU) to the main Radiology Department for imaging in an adult-sized magnetic resonance imaging (MRI) scanner. For these reasons, the smallest and/or sickest neonates are typically precluded from receiving an MRI exam. The goal of our research effort is to bring high-performance MRI into the NICU so that all neonates can benefit from the same quality of diagnostic imaging as adults. To accomplish this, we have converted a commercial small-bore 1.5 Tesla (T) MRI scanner designed for orthopedic use into a neonatal MRI system optimized for whole body imaging of neonates (NICU MRI). To expand the imaging capabilities of the NICU MRI system, the measurement control electronics and operating system software of the FDA cleared OPTIMA platform have been augmented with state of the art HDX electronics and software currently used on a conventional commercially available adult sized whole body MRI scanner. The clinical safety of the integrated HDX/OPTIMA NICU MRI system and its ability to produce diagnostic image quality has been shown in 15 pilot patients (CCHMC Protocol 2011-2045). Further we have scanned almost 600 patients under a prior protocol (CCHMC Protocol 2011-2850) without an adverse event.

The present protocol seeks to allow continued performance of clinical MRI exams on the NICU magnet with improved administrative processes and procedures. NICU patients for whom an MRI exam is medically indicated will be recruited for the present study. Images will be obtained using both the FDA cleared OPTIMA NICU MRI platform and the integrated HDX/OPTIMA NICU MRI platform with the additional HDX images augmenting the OPTIMA images and contributing to diagnosis and guidance of subsequent clinical management. The specific MR imaging methods/procedures utilized will be determined by the type of exam to be performed and the medical indication. All of the MR images obtained will be reviewed by a board certified pediatric radiologist as part of clinical care and a clinical report will be generated and included in the infant's medical record.

ELIGIBILITY:
Inclusion Criteria:

* Any infant admitted to CCHMC
* Have a medical condition for which an MRI exam is indicated, as determined by the attending neonatologist

Exclusion Criteria:

* Infants too large to fit in the customized NICU MRI system comfortably (generally infants > 6 kg)
* Standard MRI exclusion criteria as set forth by the CCHMC Division of Radiology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2018-02-11 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth M Kline-Fath, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- NICU, Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] McCormick MC, Behrman RE. The quiet epidemic of premature birth: commentary on a recent Institute of Medicine report. Ambul Pediatr. 2007 Jan-Feb;7(1):8-9. doi: 10.1016/j.ambp.2006.10.002. No abstract available. PMID 17261476
- [Background] Beck S, Wojdyla D, Say L, Betran AP, Merialdi M, Requejo JH, Rubens C, Menon R, Van Look PF. The worldwide incidence of preterm birth: a systematic review of maternal mortality and morbidity. Bull World Health Organ. 2010 Jan;88(1):31-8. doi: 10.2471/BLT.08.062554. Epub 2009 Sep 25. PMID 20428351
- [Background] Arthur R. Magnetic resonance imaging in preterm infants. Pediatr Radiol. 2006 Jul;36(7):593-607. doi: 10.1007/s00247-006-0154-x. Epub 2006 May 19. PMID 16770664
- [Background] Hirsch W, Sorge I, Krohmer S, Weber D, Meier K, Till H. MRI of the lungs in children. Eur J Radiol. 2008 Nov;68(2):278-88. doi: 10.1016/j.ejrad.2008.05.017. Epub 2008 Sep 3. PMID 18771869
- [Background] Adams EW, Counsell SJ, Hajnal JV, Allsop JM, Herlihy A, Edwards AD. Investigation of lung disease in preterm infants using magnetic resonance imaging. Biol Neonate. 2000 May;77 Suppl 1:17-20. doi: 10.1159/000047053. PMID 10828582
- [Background] Krishnamurthy R. Neonatal cardiac imaging. Pediatr Radiol. 2010 Apr;40(4):518-27. doi: 10.1007/s00247-010-1549-2. PMID 20225116
- [Background] Schweigmann G, Gassner I, Maurer K. Imaging the neonatal heart--essentials for the radiologist. Eur J Radiol. 2006 Nov;60(2):159-70. doi: 10.1016/j.ejrad.2006.07.017. Epub 2006 Aug 22. PMID 16930906
- [Background] Barkovich AJ. MR imaging of the neonatal brain. Neuroimaging Clin N Am. 2006 Feb;16(1):117-35, viii-ix. doi: 10.1016/j.nic.2005.10.003. PMID 16543088
- [Background] van Wezel-Meijler G, Leijser LM, de Bruine FT, Steggerda SJ, van der Grond J, Walther FJ. Magnetic resonance imaging of the brain in newborn infants: practical aspects. Early Hum Dev. 2009 Feb;85(2):85-92. doi: 10.1016/j.earlhumdev.2008.11.009. Epub 2009 Jan 12. PMID 19138830
- [Background] Saunders DE, Thompson C, Gunny R, Jones R, Cox T, Chong WK. Magnetic resonance imaging protocols for paediatric neuroradiology. Pediatr Radiol. 2007 Aug;37(8):789-97. doi: 10.1007/s00247-007-0462-9. Epub 2007 May 9. PMID 17487479
- [Background] Mathur AM, Neil JJ, McKinstry RC, Inder TE. Transport, monitoring, and successful brain MR imaging in unsedated neonates. Pediatr Radiol. 2008 Mar;38(3):260-4. doi: 10.1007/s00247-007-0705-9. Epub 2007 Dec 19. PMID 18175110
- [Background] Bluml S, Friedlich P, Erberich S, Wood JC, Seri I, Nelson MD Jr. MR imaging of newborns by using an MR-compatible incubator with integrated radiofrequency coils: initial experience. Radiology. 2004 May;231(2):594-601. doi: 10.1148/radiol.2312030166. PMID 15128999
- [Background] Erberich SG, Friedlich P, Seri I, Nelson MD Jr, Bluml S. Functional MRI in neonates using neonatal head coil and MR compatible incubator. Neuroimage. 2003 Oct;20(2):683-92. doi: 10.1016/S1053-8119(03)00370-7. PMID 14568444
- [Background] Foran AM, Fitzpatrick JA, Allsop J, Schmitz S, Franklin J, Pamboucas C, O'Regan D, Hajnal JV, Edwards AD. Three-tesla cardiac magnetic resonance imaging for preterm infants. Pediatrics. 2007 Jul;120(1):78-83. doi: 10.1542/peds.2006-3305. PMID 17606564
- [Background] Groves AM, Chiesa G, Durighel G, Goldring ST, Fitzpatrick JA, Uribe S, Razavi R, Hajnal JV, Edwards AD. Functional cardiac MRI in preterm and term newborns. Arch Dis Child Fetal Neonatal Ed. 2011 Mar;96(2):F86-91. doi: 10.1136/adc.2010.189142. Epub 2010 Oct 21. PMID 20971721
- [Background] Michael R. Potential of MR-imaging in the paediatric abdomen. Eur J Radiol. 2008 Nov;68(2):235-44. doi: 10.1016/j.ejrad.2008.07.017. Epub 2008 Oct 9. PMID 18848412
- [Background] Rao P. Neonatal gastrointestinal imaging. Eur J Radiol. 2006 Nov;60(2):171-86. doi: 10.1016/j.ejrad.2006.07.021. Epub 2006 Sep 25. PMID 16997526
- [Background] Riccabona M. Imaging of the neonatal genito-urinary tract. Eur J Radiol. 2006 Nov;60(2):187-98. doi: 10.1016/j.ejrad.2006.07.022. Epub 2006 Sep 7. PMID 16959460
- [Background] Darge K, Jaramillo D, Siegel MJ. Whole-body MRI in children: current status and future applications. Eur J Radiol. 2008 Nov;68(2):289-98. doi: 10.1016/j.ejrad.2008.05.018. Epub 2008 Sep 16. PMID 18799279
- [Background] Olsen OE. Practical body MRI-A paediatric perspective. Eur J Radiol. 2008 Nov;68(2):299-308. doi: 10.1016/j.ejrad.2008.06.034. Epub 2008 Sep 2. PMID 18768278
- [Background] Seghier ML, Huppi PS. The role of functional magnetic resonance imaging in the study of brain development, injury, and recovery in the newborn. Semin Perinatol. 2010 Feb;34(1):79-86. doi: 10.1053/j.semperi.2009.10.008. PMID 20109975
- [Background] Simbrunner J, Riccabona M. Imaging of the neonatal CNS. Eur J Radiol. 2006 Nov;60(2):133-51. doi: 10.1016/j.ejrad.2006.07.019. Epub 2006 Sep 14. PMID 16973325
- [Background] Rutherford M, Srinivasan L, Dyet L, Ward P, Allsop J, Counsell S, Cowan F. Magnetic resonance imaging in perinatal brain injury: clinical presentation, lesions and outcome. Pediatr Radiol. 2006 Jul;36(7):582-92. doi: 10.1007/s00247-006-0164-8. Epub 2006 May 16. PMID 16770663
- [Background] Bartha AI, Yap KR, Miller SP, Jeremy RJ, Nishimoto M, Vigneron DB, Barkovich AJ, Ferriero DM. The normal neonatal brain: MR imaging, diffusion tensor imaging, and 3D MR spectroscopy in healthy term neonates. AJNR Am J Neuroradiol. 2007 Jun-Jul;28(6):1015-21. doi: 10.3174/ajnr.A0521. PMID 17569948
- [Background] Glass HC, Bonifacio SL, Sullivan J, Rogers E, Ferriero DM, Goldstein R, Barkovich AJ. Magnetic resonance imaging and ultrasound injury in preterm infants with seizures. J Child Neurol. 2009 Sep;24(9):1105-11. doi: 10.1177/0883073809338328. PMID 19745086
- [Background] Prager A, Roychowdhury S. Magnetic resonance imaging of the neonatal brain. Indian J Pediatr. 2007 Feb;74(2):173-84. doi: 10.1007/s12098-007-0012-3. PMID 17337831
- [Background] Roelants-van Rijn AM, Groenendaal F, Beek FJ, Eken P, van Haastert IC, de Vries LS. Parenchymal brain injury in the preterm infant: comparison of cranial ultrasound, MRI and neurodevelopmental outcome. Neuropediatrics. 2001 Apr;32(2):80-9. doi: 10.1055/s-2001-13875. PMID 11414648
- [Background] Maalouf EF, Duggan PJ, Counsell SJ, Rutherford MA, Cowan F, Azzopardi D, Edwards AD. Comparison of findings on cranial ultrasound and magnetic resonance imaging in preterm infants. Pediatrics. 2001 Apr;107(4):719-27. doi: 10.1542/peds.107.4.719. PMID 11335750
- [Background] Epelman M, Daneman A, Kellenberger CJ, Aziz A, Konen O, Moineddin R, Whyte H, Blaser S. Neonatal encephalopathy: a prospective comparison of head US and MRI. Pediatr Radiol. 2010 Oct;40(10):1640-50. doi: 10.1007/s00247-010-1634-6. Epub 2010 Apr 22. PMID 20411255
- See also: Births: preliminary data for 2007. — http://www.cdc.gov/nchs/data/nvsr/nvsr57/nvsr57_12.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRI for Neonates
Started | 386
Completed | 374
Not Completed | 12
Not completed — Clinical exam moved to another scanner | 7
Not completed — Clinical order cancelled | 4
Not completed — Neonate did not settle down for the scan | 1

BASELINE CHARACTERISTICS:
Population: Neonates
Arm/Group | MRI for Neonates
Number analyzed (Participants) | 386
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 386
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: days] | 20 [1 to 155]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170
  Male | 216
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Anatomy scanned [Count of Participants; unit: Participants] — Subjects that were scheduled to complete their MRI in the NICU scanner were enrolled and the planned anatomy was documented.
  Participants
    Brain | 365
    Brain and Neonate Spine | 2
    Chest | 4
    Spine | 14
    Whole Body | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as Observed During and After Scanning.
Description: Any observed physical changes will be recorded during and after scanning
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | MRI for Neonates
Number analyzed (Participants) | 374
Participants | 0

2. Secondary Outcome: Each Infant's Baseline Measurement for Weight Will be Recorded.
Description: These measures will be used in order to facilitate future design of coils and transport tables for the customized MRI system.
Time Frame: Day 1
Measure: Mean (Full Range); unit: kg
Arm/Group | MRI for Neonates
Number analyzed (Participants) | 374
kg | 2.92 [0.54 to 4.89]

3. Secondary Outcome: Each Infant's Anatomy Scanned Will be Obtained.
Description: The anatomy used will be used in order to facilitate understand the need for specific coils for the customized MRI system.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | MRI for Neonates
Number analyzed (Participants) | 374
Participants
  Brain | 357
  Brain and Neonate Spine | 1
  Chest | 2
  Spine | 13
  Whole Body | 1

4. Secondary Outcome: Baseline Measurement for Days Old Will be Recorded.
Description: These measures will be used in conjunction with the weight at the time of scan to facilitate future design of coils and transport tables for the customized MRI system.
Time Frame: Day 1
Measure: Median (Full Range); unit: days
Arm/Group | MRI for Neonates
Number analyzed (Participants) | 386
days | 20 [1 to 155]

ADVERSE EVENTS:
Time Frame: Time that participant was in the NICU scanner for their clinically indicated scan (length of scan varies based on standard of care exam).
Arm/Group | MRI for Neonates
All-Cause Mortality (participants affected / at risk) | 0/374
Serious Adverse Events (participants affected / at risk) | 0/374
Other Adverse Events (participants affected / at risk) | 0/374

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT03476343/Prot_001.pdf